CLINICAL TRIAL: NCT06257303
Title: Investigation of the Correlation Between Dynamic Knee Valgus and Landing Biomechanics, Core Endurance and Ankle Dorsiflexion in Adolescent Female Basketball Players
Brief Title: Relationship Between Knee Valgus and Landing Biomechanics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bahçeşehir University (Other)
Responsible Party: Principal Investigator, Pelin Pişirici, Assistant Professor, PT, PhD, Bahçeşehir University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NA-LandingB
Record Dates: First submitted 2024-02-05; First posted 2024-02-13 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Injury Traumatic; Injury;Sports; Injury, Knee; Injury, Ankle
Keywords: injury preventation; frontal plane projection angle; landing error scoring system; weight bearing lunge test
MeSH Terms: conditions — Wounds and Injuries; Athletic Injuries; Knee Injuries; Ankle Injuries

STUDY DESIGN:
Intervention Model Description: Participants will be divided into two groups according to the presence of frontal plane projection angle and their demographic characteristics will be compared.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be blinded to the purpose of the study. In this way, it is planned to prevent them from making corrections in their alignment or posture.
  The evaluator will also be blind to the groups. After the frontal plane projection angle measurement, it will be determined which group the participant will be in. Still, this information will not be shared with the evaluator who makes other evaluations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Valgus Group (Active Comparator): If there is an increase of 10 degrees or more in the frontal plane projection angle while squatting on one leg, the participant will be included in this group.
  Interventions: Other: Frontal Plane Projection Angle
- Control Group (Active Comparator): If the frontal plane projection angle is in the normal values while squatting on one leg, the participant will be included in this group.
  Interventions: Other: Frontal Plane Projection Angle

INTERVENTIONS:
Other: Frontal Plane Projection Angle — Participants will stand with their feet aligned in the sagittal plane and their arms crossed across their chests. By prior instruction, subjects will be asked to squat up to 60º knee flexion in a controlled manner without losing their balance, before returning to the starting position. Digital recordings of the frontal plane will be made while individuals perform a single-leg squat test at 60º knee flexion 3 times.

SUMMARY:
It has been shown that especially adolescent female athletes have a very high risk of injury compared to males. Gender differences (anatomical, biomechanical, neuromuscular and hormonal differences) contribute to the increased risk of injury. Basketball, one of the sports preferred by adolescent girls, brings with it high risks of injury due to the high participation rate among team sports. The occurrence of lower extremity injuries such as anterior cruciate ligament injuries and patellofemoral pain during dynamic activities (e.g., landing, running, etc.) has been associated with dynamic knee valgus, a pattern of lower extremity malalignment. At the same time, weakness of the core muscles and inadequate ankle dorsiflexion joint range of motion also contribute to the injury. The aim of this study is to examine the correlation between landing biomechanics, core endurance and ankle dorsiflexion angle in adolescent female basketball players with dynamic knee valgus.

DETAILED DESCRIPTION:
Although interest in identifying injury risk factors has increased recently, it has been stated that adolescent athletes are especially vulnerable to injury. Such sex-based differences that may explain the increased risk of anterior cruciate ligament injury in girls compared with boys include anatomical, biomechanical, neuromuscular, and hormonal differences. A broad range of physiological mechanisms (e.g., hormone control, differences in joint geometry, collagen turnover, etc.) play a role in lower extremity injuries and may explain these sex differences. Basketball, one of the sports preferred by adolescent girls, brings with it high risks of injury due to the high participation rate among team sports. As a result of the studies, it was revealed that 7 to 10 people out of every 1000 were injured. 16% of female basketball players are at risk of anterior cruciate ligament injury during their careers, and this rate is 2 to 4 times higher than that of men. The occurrence of lower extremity injuries such as anterior cruciate ligament injuries and patellofemoral pain during dynamic activities (e.g., landing, running, etc.) has been associated with dynamic knee valgus. A common malalignment that may occur in the lower extremities during sports activities is dynamic knee valgus, which has been suggested as the underlying mechanism of knee injury. Dynamic knee valgus involves a combination of knee abduction, tibial internal rotation, and hip adduction. Numerous studies associate core muscle weakness with lower extremity malalignment. Changes in the trunk-pelvis-hip complex can lead to dynamic knee valgus, a dysfunction that also appears to be influenced by factors such as gender, physical activity level, and body mass index. In post-jump landing biomechanics, limitations in ankle dorsiflexion joint range of motion are considered a modifiable injury risk factor for athletes. Ankle dorsiflexion during landing helps reduce ground reaction forces and facilitates knee and hip flexion in the sagittal plane. It has been shown that decreased ankle dorsiflexion joint range of motion limits peak flexion angles of the ankle, knee, and hip and increases peak knee abduction angles during descent. This situation shows the relationship between ankle dorsiflexion joint range of motion and frontal plane projection angle. This study aims to examine the correlation between landing biomechanics, core endurance and ankle dorsiflexion angle in adolescent female basketball players with dynamic knee valgus. It was hypothesized that participants with greater knee valgus had poor core stabilization ability and limited dorsiflexion angle.

ELIGIBILITY:
Inclusion Criteria:

* Having been training basketbol for at least 6 months,
* Being between the ages of 10-19
* Being female
* Having an increase of 10 degrees or more in the frontal plane projection angle (for the valgus group)
* Having a frontal plane projection angle at normal values (for the control group)
* No active pain in the lower extremity
* No mental and psychological problems

Exclusion Criteria:

* Non-volunteer athletes
* Having a body mass index of 30 kg/m² and above
* Having undergone lower extremity surgery
* Having chronic knee instability.
* Having had a meniscus or ligament injury
* Having a cardiac, musculoskeletal, vestibular and neurological disease
* Having been using corticosteroids and nonsteroidal drugs for a long time.
* Being pregnant.

Ages: 10 Years to 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 56 (Actual)
Dates: Start 2024-04-30 (Actual); Primary Completion 2025-01-10 (Actual); Study Completion 2025-01-10 (Actual)

PRIMARY OUTCOMES:
Landing Error Scoring System | Baseline
  The Landing Error Scoring System (LESS) is a screening tool used to identify athletes who exhibit movement patterns that pose a high risk of injury in post-jump landing biomechanics. Evaluaters will score 17 items based on movements during the jump-landing task. The overall LESS score ranges from 0 to 17 errors, with lower scores reflecting fewer landing errors. An error score of five or more indicates poor jumping technique and is associated with a higher risk of lower extremity injury. Participants will begin LESS standing on a 30 cm high box and will be asked to jump forward a distance equal to half their height (indicated by a line on the ground) and make a maximum vertical jump once they land. Participants will be provided with a verbal explanation and visual demonstration before testing and will be allowed to try the procedure until they become familiar with it. Each participant will complete 3 trials of LESS and the resulting average will be considered for analysis.

SECONDARY OUTCOMES:
Core endurance assessment tests | Baseline
  The prone plank test will be used to evaluate trunk flexor endurance. For the prone plank test, participants will maintain a prone position in which their body weight is supported by the toes and forearms.
  The side plank test will be performed with the participant lying on their side, supported by their foot and elbow. The side plank test will be performed on both sides. Participants will be instructed to maintain a neutral position of the spine and pelvis and breathe normally during the test. Each test will be terminated when the participant is unable to maintain posture or their pelvis moves up or down five or more cm. Each hold time will be recorded using a stopwatch.
  When 1 minute is completed in both tests, chorea muscle strength will be considered sufficient.
Weight-bearing lunge test | Baseline
  Weight-bearing lunge test (WBLT) is frequently used in individuals with ankle instability to determine dorsiflexion normal joint movement. During WBLT the participant puts his hands on the wall and takes one leg forward and the other leg helps balance behind. The maximum distance that the knee touches the wall is recorded without allowing the heel of the front foot to lose contact with the ground. The clinically significant value for WBLT was determined as 2.5 cm.

CONTACTS AND LOCATIONS:
Locations (1):
- Bahcesehir University, Istanbul, Turkey (Türkiye)